CLINICAL TRIAL: NCT01018368
Title: An Open-Label Phase 1 Study to Examine the Effect of Multiple Doses of Rifampin on the Single-Dose Pharmacokinetics of VX 770 in Healthy Subjects
Brief Title: Study of VX-770 and Rifampin in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Medical Monitor, Vertex Pharmaceutical Incorporated
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VX09-770-009
Record Dates: First submitted 2009-11-19; First posted 2009-11-23 (Estimated); Last update posted 2010-05-10 (Estimated); Status verified 2010-05

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VX-770 (Experimental)
  Interventions: Drug: VX-770
- Rifampin (Experimental)
  Interventions: Drug: Rifampin

INTERVENTIONS:
Drug: VX-770 — In Period 1, subjects will receive a single oral dose of VX-770 150 mg on Day 1. In Period 2, subjects will receive a single oral dose of VX-770 150 mg on Day 6.
  Arms: VX-770
Drug: Rifampin — In Period 2, subjects will receive a daily oral dose of rifampin 600 mg on Days 1 through 10
  Arms: Rifampin

SUMMARY:
The objectives of this study are to evaluate the effects of multiple doses of rifampin on the single-dose pharmacokinetics of VX 770.

DETAILED DESCRIPTION:
This is a single-center, nonrandomized, open-label, 2-period, 1-sequence crossover study to investigate the safety, tolerability and pharmacokinetics of VX 770 when administered alone or with rifampin.

All enrolled subjects will receive the same treatments and undergo the same procedures. In Period 1, subjects will receive a single dose of VX 770 on Day 1. In Period 2, subjects will receive a daily dose of rifampin on Days 1 through 10 and a single dose of VX 770 on Day 6.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be male and between 18 and 55 years of age
* Subject must have a body mass index (BMI) from 18 to 30 kg/m2

Exclusion Criteria:

* History of any illness or condition that, in the opinion of the investigator might confound the results of the study or pose an additional risk in administering study drug to the subject
* Subjects who have active tuberculosis, human immunodeficiency virus, hepatitis C, or active hepatitis B

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
VX 770 pharmacokinetic (PK) parameters | 17 days

SECONDARY OUTCOMES:
VX 770 metabolite PK parameters in plasma | 17 days
Rifampin concentration at time zero (C0) and AUC at steady state (AUCtau) following the administration of multiple doses of rifampin | 17 days
Safety as measured by adverse events, physical examinations, vital signs, electrocardiograms (ECGs), and clinically significant laboratory assessments | 17 days

CONTACTS AND LOCATIONS:
Overall Officials: H. Frank Farmer, MD, Principal Investigator — Covance CRU, Inc.
Locations (1):
- Daytona Beach, Florida, United States